CLINICAL TRIAL: NCT06130917
Title: Effects of Multisystem Exercise Program on Balance, Postural Stability, Mobility and Pain in Patients With Diabetic Peripheral Neuropathy
Brief Title: Effects of Multisystem Exercise on Balance, Postural Stability, Mobility and Pain in Patients With DPN.
Acronym: DPN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/0242 Sidra khurshid
Record Dates: First submitted 2023-11-09; First posted 2023-11-14 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Diabetic Peripheral Neuropathy
Keywords: Balance, Multisystem Exercise, Peripheral neuropathy
MeSH Terms: conditions — Peripheral Nervous System Diseases | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and outcome assessors will be kept blinded about the intervention which the patients will be going to receive.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Experimental group will receive education on diabetes and conventional treatment exercises. The interventional multisystem exercises program will consist of four components, with each exercise lasting for a duration of 10 minutes per session. These components encompass proprioception training, balance exercises, strengthening routines, and reaction time training. This total multisystem exercises session will be performed for 30 minute, 3 times a week for 8 weeks in total.
  Interventions: Other: Multisystem Exercise
- Control group (Other): Control group will receive health education on diabetes. Conventional treatment will include Stretching, Range of motion (ROM) exercise , balance and strengthening for 10 minutes each exercise in one session. Each stretch holds for 15-20 sec. This exercise session will be performed for 30 minute, 3 times a week for 8 weeks in total.
  Interventions: Other: Conventional Treatment

INTERVENTIONS:
Other: Multisystem Exercise — Proprioception: Seated ankle ball. Single leg stance with support and with extension of knees. Single leg stance (hip extension) with support and with extension' of knees.
  Muscle strengthening: Seated alternate double knee lifts with weights, chair stands. Seated alternate kicks with weigh. Hip extension standing with support with weights.
  Balance Training Seated alternate weight shifts. Seated calf and toe raise. Heel raise with support.. Crossover with support Reaction time Seated alternate touches to front. Seated alternate touches to back. Seated alternate touches to side. Seated alternate touches to 3 steps (forward, side, backward).
  Other Names: Experimental Group
  Arms: Experimental Group
Other: Conventional Treatment — ROM exercises Passive ROM exercise of hip. Passive ROM exercise of knee. Passive ROM exercise of ankle Muscle strengthening Seated alternate double knee lifts with weights. chair stands. Seated alternate kicks with weigh. Hip extension standing with support with weights.
  Balance Seated alternate weight shifts. Seated calf and toe raise. Heel raise with support. Crossover with support Stretching exercises Stretching exercise of hamstring. Stretching exercise of quadriceps. Stretching exercise of calf muscle
  Other Names: Control Group
  Arms: Control group

SUMMARY:
Upto the best knowledge of researcher, multisystem exercise program has been utilized in various populations, encompassing both healthy individuals and patients with diverse medical conditions. However, its specific impact on the diabetic peripheral neuropathy population, particularly in terms of improving balance, postural stability and mobility remains inadequately explored.

DETAILED DESCRIPTION:
Diabetic peripheral neuropathy is a common and highly prevalent complication of type 2 diabetes mellitus, posing a significant global health concern. It affects a considerable number of individuals with diabetes, leading to progressive nerve damage and functional impairments. The multifaceted nature of this condition manifests in various ways, including sensory, motor, and autonomic dysfunction. Its insidious onset and gradual progression impose a substantial burden on patients, reducing their quality of life and presenting significant challenges for healthcare providers. Therefore, understanding the underlying causes, mechanisms, and management strategies of diabetic peripheral neuropathy is essential to alleviate its impact and enhance the overall well-being of those affected by this condition. Patients with diabetic peripheral neuropathy encounter a range of distressing symptoms that profoundly influence their daily activities. Sensory manifestations, such as numbness, tingling, and pain, are common, especially among older individuals with diabetes. Challenges in detecting temperature and touch also increase the risk of burns or injuries. Motor neuropathy results in muscle weakness, loss of balance, and coordination difficulties, making simple tasks like walking or holding objects more challenging. Furthermore, diabetic peripheral neuropathy plays a significant role in falls among elderly patients due to balance disorders and proprioception impairment. To address these issues and improve patients' quality of life, exercise has emerged as a valuable therapeutic intervention. Regular exercise programs, specifically those incorporating balance training exercises, have shown promising outcomes in enhancing balance and reducing falls among those with diabetic peripheral neuropathy. By emphasizing a comprehensive approach to exercise, targeting proprioception, coordination, and lower limb strength, patients can benefit from improved sensory integration, enhanced muscle control, and postural stability, ultimately promoting greater independence and reducing the risk of falls. Through a well-designed randomized controlled trial, exploring the effectiveness of a multisystem exercise program, further advancements in managing diabetic peripheral neuropathy can be achieved, leading to improved patient outcomes and enhanced quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Both genders (male, female)
* Age (40-60)
* Patients who are screened for diabetic peripheral neuropathy
* Moderate balance impairment on Berg Balance Scale (21-40)
* Patients who met the criteria of Diabetic Neuropathy 4 scored equal or greater than 4.
* Patients who have positive sharpened Romberg test

Exclusion Criteria:

* Patients with any recent surgery of lower limb
* Patients with crutches
* Patients with gangrene
* Patients with lower BMI
* patients with Deep Venous Thrombosis (DVT)
* patients with amputations
* Patients with neurological impairments in the central nervous system and vestibular system
* Patients with orthostatic hypotension

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2023-11-05 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2024-04-10 (Actual)

PRIMARY OUTCOMES:
Beg Balance Scale | 8 weeks
  It is used to assess balance. Each item is a 5-point ordinal scale ranging from 0 to 4, with 0 indicating an inability to complete the task entirely and 4 indicating an ability to complete the task criterion. Scores can range from 0 to 56. Change will be measured from Baseline to 8 weeks.
Functional reach test | 8 weeks
  It is a widely used clinical assessment tool to measure an individual's dynamic balance and stability. The test requires the participant to reach forward as far as possible without taking a step or losing balance. The distance reached is recorded and compared to normative values based on age and gender. score less than 6 indicates risk of fall. score between 6-10 indicates moderate risk of fall. Change will be measured from baseline to 8 weeks
Timed Up and Go test | 8 weeks
  It is for the assessment of lower extremity function, mobility and fall risk. score more than 12 indicates risk of fall and walking problem. Change will be measured from Baseline to 8 weeks.
Ten meter walk test | 8 weeks
  It is a performance measure used to assess walking speed in meters per second over a short distance. its value for adults between 40 to 60 ages ranges from 1.43 to 1.31 m/s. Change will be measured from Baseline to 8 weeks
Numeric pain rating scale | 8 weeks
  Numeric Pain Rating Scale (NPRS) is used to assess the pain levels reported by participants. it ranges from 0 to 10, with 0 indicating no pain and 10 representing the most awful imaginable pain. Change will be measured from Baseline to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Aruba Saeed, PhD*, Principal Investigator — Riphah International University Pakistan
Locations (1):
- DHQ Pakpattan, Pakpattan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khurshid S, Saeed A, Kashif M, Nasreen A, Riaz H. Effects of multisystem exercises on balance, postural stability, mobility, walking speed, and pain in patients with diabetic peripheral neuropathy: a randomized controlled trial. BMC Neurosci. 2025 Feb 27;26(1):16. doi: 10.1186/s12868-024-00924-6. PMID 40016658